CLINICAL TRIAL: NCT05720975
Title: First Prospective, Single-arm, Single-centre Study to Evaluate the Efficacy and Safety of the Thromboaspiration Catheter System (iNstroke) for Stroke in Patients With Acute Ischemic Stroke
Brief Title: Efficacy and Safety Evaluation of the Thromboaspiration Catheter System iNstroke in Patients With Acute Ischemic Stroke
Acronym: ASPiC
Status: Completed | Type: Observational
Sponsor: iVascular S.L.U. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASPiC-01
Record Dates: First submitted 2022-07-21; First posted 2023-02-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Ischemia; Thromboaspiration
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental: iNstroke: Study device
  Interventions: Device: iNstroke

INTERVENTIONS:
Device: iNstroke — Patients to undergo thromboaspiration with iNstroke.

SUMMARY:
First prospective, single-arm, single-centre study to evaluate the efficacy and safety of the iNstroke thromboaspiration catheter system (iNstroke) for stroke in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-centre clinical safety and efficacy research.

The purpose of the study is to evaluate safety and efficacy the device designed by iVascular for thromboaspiration (iNstroke) in patients who have suffered a stroke and who undergo thromboaspiration due to an acute occlusion of neuro vessels.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute ischaemic stroke over 18 years of age caused by large vessel occlusion (TICA, extracranial ICA, M1, vertebral artery segment V4 or basilar artery) and receiving neurointerventional treatment with the iNstroke aspiration catheter.
2. Informed consent signed by the patient or their representative, or deferred informed consent to avoid delaying commencement of mechanical thrombectomy.
3. Patients with an ASPECTS (Alberta Stroke Program Early CT Score) score ≥ 6
4. In patients having onset of stroke more than 8 hours previously, wake-up strokes, or unknown time of onset, treatment must be customised and CT perfusion must show penumbra.
5. Initial NIHSS score before procedure > 6.

Exclusion Criteria:

1. Patients under 18 years of age.
2. Patients with an ASPECTS score <6.
3. Baseline NIHSS obtained before procedure of ≤ 6 points.
4. Severe comorbidity and/or shortened life expectancy
5. mRS > 2.
6. Serious allergy to contrast medium.
7. Pregnant women.
8. Patients with intracranial atherosclerotic occlusive disease or extra- or intracranial dissection
9. Personal history of thrombocytopaenia (<40,000 platelets)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients experiencing acute ischaemic stroke of the anterior circulation with occlusion of TICA, M1, extracranial ICA, vertebral artery segment V4 or basilar artery, treated with iNstroke aspiration catheter and complying with the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Performance success | In the course of cervico-cranial catheterization, evaluated immediately after endovascular procedure.
  Recanalization rate with mTICI ≥2b-3 (modified thrombolysis in cerebral infarction scale).
MAE | 24 hours (-8/+12 hours)
  All serious adverse events.
Mortality | 90 days
  All-cause mortality.

SECONDARY OUTCOMES:
Navigability | In the course of cervico-cranial catheterization, evaluated immediately after endovascular procedure.
  Number of procedures in which the InStroke catheter reaches the intracranial occluded segment (M1, basilar artery) through coaxial system with a microcatheter and without the assistance of other additional devices.
Clinical progress | 90 days
  Good functional clinical progress (modified Rankin scale 0-2).
Proportion of patients with rapid neurological improvement | 24 hours
  Proportion of patients with rapid neurological improvement (more than 4 points on the NIHSS scale)
Reduction of NIHSS scale | 24 or 72 hours
  Proportion of patients with a reduction of ≥8 points on the NIHSS scale (during the first 24 hours post-treatment), or NIHSS 0-1 (at 72 hours [or at the time of discharge, whichever occurs first]).
Procedure duration | In the course of cervico-cranial catheterization, evaluated immediately after endovascular procedure.
  Procedure duration defined as the time from puncture to when grade ≥2b is reached on the mTICI scale with less than three passes or, if not achieved, until the final angiogram.
Number of passes with the device until recanalisation. | In the course of cervico-cranial catheterization, evaluated immediately after endovascular procedure.
  Number of passes with the device until recanalisation.
Percentage of effective recanalisation in a first pass | In the course of cervico-cranial catheterization, evaluated immediately after endovascular procedure.
  Percentage of effective recanalisation in a first pass, the effect of which will be measured by a recanalisation rate of TICI2c-3 and TICI 2b-3.
Rate of need to use another reperfusion technique | In the course of cervico-cranial catheterization, evaluated immediately after endovascular procedure.
  Rate of need to use another reperfusion technique due to suction system failure.
Assessment of symptomatic intracerebral haemorrhage | 24 (-8/+12) hours.
  Assessment of symptomatic intracerebral haemorrhage by magnetic resonance imaging (MRI)/computed tomography (CT). ICH is defined as the presence of extravascular blood in the brain or within the skull- ICH is considered symptomatic (SICH) if it is associated with clinical deterioration (worsening of the score National Institutes of Health Stroke Scale (NIHSS) of
  ≥4 points) or if it causes death and is identified as the predominant cause of neurological deterioration, according to the assessment of an independent clinical events committee (CEC).
Neurological deterioration | 24 (-8/+12) hours.
  Classification of neurological deterioration of ≥4 points on the NIHSS scale.
Embolization rate | In the course of cervico-cranial catheterization, evaluated immediately after endovascular procedure.
  Embolization rate in a previously non-involved territory on cerebral angiography.
Mortality rate | 3 days (+/-24 hours) or at discharge, whichever occurs first.
  Mortality rate related to the procedure
Procedure complication rate | In the course of cervico-cranial catheterization, evaluated immediately after endovascular procedure.
  Procedure complication rate: arterial perforation, arterial dissection and severe vasospasm in the target vessel

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: No